CLINICAL TRIAL: NCT01427075
Title: Evaluation of the Pharynx Through MRI in Patients Undergoing Lateral Pharyngoplasty for Treatment of Obstructive Sleep Apnea
Brief Title: Evaluation Of The Pharynx in Patients Undergoing Lateral Pharyngoplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital do Servidor Publico Estadual (Other)
Responsible Party: Principal Investigator, CAROLINA DE ANDRADE FERREIRA VIEIRA, VIEIRA, CAF, Hospital do Servidor Publico Estadual
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 018/11
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Magnetic Resonance Imaging; Sleep Apnea, Obstructive; Pharyngeal Muscles
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lateral pharyngoplasty (Experimental): lateral pharyngoplasty
  Interventions: Procedure: LATERAL PHARYNGOPLASTY

INTERVENTIONS:
Procedure: LATERAL PHARYNGOPLASTY — tonsilectomy and lateral pharyngoplasty

SUMMARY:
This study will evaluate the pharynx in patients undergoing lateral pharyngoplasty for treatment of obstructive sleep apnea through MRI, before and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of obstructive sleep apnea syndrome

Exclusion Criteria:

* MRI contraindications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
expansion of pharynx | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: CAROLINA AF VIEIRA, MD, Principal Investigator — Hospital do Servidor Publico Estadual
Locations (1):
- Hospital Do Servidor Publico Estadual, São Paulo, São Paulo, Brazil